CLINICAL TRIAL: NCT05456178
Title: Evaluation of the Relationship Between the Degree of Environmental Fungal Exposure in Patients' Dwellings and Clinical Symptoms of Patients With Chronic Obstructive Pulmonary Disease - Study of Feasibility
Brief Title: Relationship Between Degree of Domestic Environmental Fungal Exposure and Clinical Symptoms of Patients With Chronic Obstructive Pulmonary Disease
Acronym: BPCO-Myc
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0913
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; Pulmonary aspergillosis; environmental fungal exposure; electrostatic wipe
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 blood sample of 3.5 ml for:
  * aspergillosis serology (Aspergillus IgG, total IgE and specific IgE for Cladosporium, Alternaria, Penicillium, Botritis, Fusarium, Candida, Schizophyllum, Curvularia, Bipolaris
  * Blood count
  One sample of expectoration for fungal diversity analysis
  An electrostatic wipe will be left in the living room and another one in the bedroom for 12 weeks. The wipes will be analyzed by the mycology laboratory of the Croix Rousse hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult subjects with chronic obstructive pulmonary disease: In adult patients with chronic obstructive pulmonary disease, an electrostatic wipe will be deposited in the living room and another one in the bedroom for 12 weeks, to be analyzed by the mycology laboratory of the Croix-Rousse hospital, Lyon.
  Interventions: Other: Electrostatic wipe

INTERVENTIONS:
Other: Electrostatic wipe — The main objective will be to study the feasibility of the quantification of domestic fungal exposure with electrostatic wipe. The interval of environmental fungal exposure quantification values measured by conventional mycology and by NGS will be established, with analysis of the correlation between the quantification obtained by the two techniques.
  For this, an electrostatic wipe will be deposited in the living room and another one in the bedroom for 12 weeks. The wipes will be analyzed by the mycology laboratory of the Croix Rousse hospital.

SUMMARY:
Exposure to Aspergillus spores is associated with symptoms of asthma or airway inflammation (Chaudhary & Marr, 2011; Smith & Denning, 2011), leading to the possible onset of severe fungal complications with acute or chronic inflammation. In patients with chronic obstructive pulmonary disease (COPD), whose main etiological factor is cigarette smoke, A. fumigatus sensitization has been reported to be related to poor lung function (Bafadhel et al., 2014). Besides, COPD patients with fungal sensitization exhibit greater granulocyte count, implying more severe inflammation (Agarwal, Gaur, & Chowdhary, 2015). Fungal cultures from sputum are frequently positive in patients with asthma or with COPD (Pashley, 2014). Fungal colonization and infection have also been suspected to be related to exacerbations of COPD, but their potential role in the pathogenesis of COPD is poorly understood (Bafadhel et al., 2014). The hypothesis is that patients with COPD have a worsening of their pulmonary symptoms after exposure to fungal spores. This study will ensure the feasibility of quantifying environmental fungal exposure in patients' dwellings. For this, an electrostatic wipe will be deposited in the living room and another one in the bedroom for 12 weeks. The wipes will be analyzed by the mycology laboratory of the Croix Rousse hospital.

If the results of this first study are conclusive, it is planned to continue this analysis with a regional multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 40
* Suffering from COPD (chronic obstructive pulmonary disease), diagnosed by a pulmonologist
* Presence of bronchial obstruction with FEV1 (Forced expiratory volume)/FVC (Forced vital capacity) <70%
* FEV reversibility post β2-mimetic < 12% and < 200 ml (vs FEV prebronchodilator)
* Smoking ≥ 10 PA active or not
* Occupied the same residence for at least 12 months
* No changes to the home or recent work in the 6 months preceding inclusion
* Delivery of enlightened information and collection of non-opposition

Exclusion Criteria:

* Other chronic respiratory diseases: asthma, bronchiectasis,
* bronchial cancer, pulmonary fibrosis, diseases requiring the use of immunosuppressive treatment or biotherapy, or any long-term treatment with oral corticosteroids used for the treatment of a disease other than COPD
* COPD exacerbation of less than 4 weeks
* Treatment with inhaled corticosteroids alone,
* Long-term treatment with oral corticosteroids
* Persons deprived of liberty by a judicial or administrative decision,
* people undergoing psychiatric care, people admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure
* Patient enrolled in interventional research excluding routine care research (former regulations) and category 2 research that does not interfere with the analysis of the primary endpoint

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns adult subjects with chronic obstructive pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Quantification of domestic fungal exposure. | 12 weeks after inclusion.
  The main judgment criterion will be to study the feasibility of the quantification of domestic fungal exposure.
  Fungal diversity exposure will be analyzed by mycological culture and next-generation sequencing.
  The interval of environmental fungal exposure quantification values measured by conventional mycology and by Next Generation Sequençing will be established, with analysis of the correlation between the quantification obtained by the two techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Jean MENOTTI, MD, Principal Investigator — Service de Parasitologie et Mycologie médicale / Institut des Agents Infectieux
Locations (1):
- Service de Parasitologie et Mycologie médicale / Institut des Agents Infectieux, Hôpital de la Croix-Rousse, HCL, Lyon, France